CLINICAL TRIAL: NCT00014261
Title: A Phase-I Study Of Cyclical Oral Administration Of Temozolomide In Combination With PEG12000-Interferon Alfa-2B In Patients With Refractory And/Or Advanced Solid Tumors
Brief Title: Temozolomide Plus PEG-Interferon Alfa-2B in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Lionel.D.Lewis, MD, Professor of Medicine and of Pharmacology and Toxicology, Dartmouth-Hitchcock Medical Center
Purpose: Treatment
Other Study IDs: CDR0000068523; P30CA023108 (NIH); DMS-0010; NCI-G01-1924
Record Dates: First submitted 2001-04-10; First posted 2003-07-30 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — peginterferon alfa-2b; Temozolomide

INTERVENTIONS:
Biological: PEG-interferon alfa-2b
Drug: temozolomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. PEG-interferon alfa-2B may interfere with the growth of cancer cells. Combining temozolomide with PEG-interferon alfa-2B may be an effective treatment for advanced solid tumors.

PURPOSE: Phase I trial to study the effectiveness of combining temozolomide and PEG-interferon alfa-2B in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and tolerability of temozolomide and PEG-interferon alfa-2b in patients with advanced refractory solid tumors or chemotherapy-naive advanced cancer.
* Determine the maximum tolerated dose (MTD) and dose-limiting toxicity of this regimen in this patient population.
* Determine the pharmacokinetics of PEG-interferon alfa-2b at the MTD when administered with temozolomide in this patient population.
* Determine the anti-tumor activity of this regimen in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive oral temozolomide on days 1-7 and 15-21 and PEG-interferon alfa-2b subcutaneously on days 1, 8, 15, and 22. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 1-9 patients receive escalating doses of temozolomide and PEG-interferon alfa-2b until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A maximum of 24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced solid tumor that is refractory to standard therapy OR
* Histologically confirmed chemotherapy-naive advanced cancer for which no curative therapy or higher priority palliative chemotherapy exists
* Brain metastasis allowed
* No bone marrow involvement of tumor

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count greater than 1,500/mm^3 AND/OR
* Platelet count greater than 100,000/mm^3

Hepatic:

* ALT or AST less than 3 times upper limit of normal (ULN) (5 times ULN if liver metastases present)
* No autoimmune hepatitis

Renal:

* Creatinine less than 2.5 times ULN

Cardiovascular:

* No severe coronary artery disease
* No congestive heart failure

Pulmonary:

* No severe chronic obstructive pulmonary disease

Gastrointestinal:

* No frequent vomiting
* No medical condition that would interfere with oral medication intake (e.g., partial bowel obstruction, partial intestinal bypass, or external biliary diversion)

Other:

* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No known or suspected hypersensitivity to imidazotetrazin, interferon alfa, or any excipient or vehicle included in the formulation or delivery system of study drug
* No history of autoimmune disease
* No preexisting severe psychiatric condition or history of severe psychiatric disorder (including suicidal ideation or attempt)
* No life-threatening condition or severe preexisting condition
* No uncontrolled thyroid abnormalities
* No nonmalignant systemic disease
* No active uncontrolled infection
* HIV negative
* No AIDS-related illness
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 3 weeks since prior biologic agents (e.g., bi-specific antibodies, interleukin-2, or interferon) and recovered (excluding alopecia)
* No prior allogeneic, syngeneic, or autologous bone marrow or stem cell transplantation
* No other concurrent biologic therapy
* No concurrent colony stimulating factors or epoetin alfa for the prevention of myelotoxicity

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy (more than 6 weeks for nitrosoureas, melphalan, or mitomycin) and recovered (excluding alopecia)
* No prior high-dose chemotherapy and stem cell transplantation
* No more than 3 prior chemotherapy regimens
* No other concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 6 weeks since prior wide-field radiotherapy to at least 25% of bone marrow (e.g., pelvic radiotherapy)
* More than 6 weeks since prior strontium chloride Sr 89 or samarium Sm 153 lexidronam pentasodium
* Recovered from prior radiotherapy (excluding alopecia)
* No concurrent radiotherapy

Surgery:

* At least 4 weeks since prior major surgery
* At least 1 week since prior minor surgery

Other:

* At least 4 weeks since prior investigational therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-10 (Actual); Primary Completion 2002-11 (Actual); Study Completion 2002-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lionel D. Lewis, MD, Study Chair — Norris Cotton Cancer Center
Locations (1):
- Norris Cotton Cancer Center, Lebanon, New Hampshire, United States